CLINICAL TRIAL: NCT02303067
Title: Prospective International Study of Coronary Subtraction Using 320 Row-Detector CT
Brief Title: Prospective International Study of Coronary Subtraction Using 320 Detector Row CT (CorSub)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150026; 15-H-0026
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2018-08-13

CONDITIONS: Coronary Artery Disease
Keywords: Cardiac; Computed Tomography; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Background:

- This study is designed for people who need a standard, non-research invasive coronary angiogram to find out if they have heart disease. Researchers want to take a computed tomography (CT) scan of people s hearts before their procedure to see if this less invasive test can also diagnose coronary artery disease.

Objectives:

- To learn if a new way to view CT pictures is able to accurately diagnose coronary artery disease.

Eligibility:

- People age 55 and older who need a coronary angiogram.

Design:

* Participants will be screened with their medical records.
* Participants may give a blood sample.
* Participants may have a CT scan of the heart with and without contrast. The CT scan will not interfere with their medical care.
* Participants blood pressure and heart rhythm will be monitored before, during, and after the CT scan. They may have an electrocardiogram.
* Before the scan, participants will have an intravenous catheter put into their arm. It will be used to inject contrast.
* Participants may take a beta blocker to slow their heart rate.
* Participants may take nitroglycerin under their tongue. It will enlarge their heart blood vessels and improve picture quality. It may cause a flushing sensation or headache.
* Participants will lie on their back on a padded table. The table slides into a large, donut-shaped machine. An x-ray tube will move around their body, taking pictures. They will be asked to hold their breath for 5 seconds at a time.
* Participants will be called 30 days after their angiogram. They will answer questions about their health, hospital visits, or medical treatments.

DETAILED DESCRIPTION:
Coronary calcium can impair the accurate evaluation of the coronary arteries with coronary computed tomography angiography (CCTA). A novel approach to potentially overcome this limitation is coronary calcium subtraction, where areas of calcification identified on a non-contrast scan are removed from the contrast enhanced images.

.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age over 55 years
  2. Subjects referred for coronary angiography
  3. Able to understand and willing to sign the Informed Consent Form

EXCLUSION CRITERIA:

1. Known allergy to iodinated contrast media
2. Estimated GFR less than 50 ml/min
3. Atrial fibrillation or other continuous cardiac arrhythmias
4. Known or suspected intolerance or contraindication to beta-blocker medication (i.e. significant reactive airway disease, decompensated heart failure, Mobitz type 2 second degree or 3rd degree atrio-ventricular heart block)
5. Inability to adequately hold breath for 5 seconds
6. Pregnancy. Women of child bearing potential must demonstrate a negative pregnancy test within 24 hours of the study MDCT.

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-01-06; Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Coronary substraction CCTA improves the diagnostic accuracy. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Y Chen, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Rigshospitalet, Copenhagen, Denmark